CLINICAL TRIAL: NCT06512883
Title: Phase 3, Open-label Trial to Evaluate Safety, Pharmacokinetics, and Efficacy of Benralizumab in Children With Eosinophilic Diseases (CLIPS)
Brief Title: A Trial to Investigate Benralizumab in Children With Eosinophilic Diseases
Acronym: CLIPS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3255C00004; 2023-508533-14-00 (Other: EU CT); EMEA-001214-PIP09-21-M02(EGPA) (Other: Paediatric Investigational Plan Number); EMEA-001214-PIP04-19-M02 (HES) (Other: Paediatric Investigational Plan Number)
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Eosinophilic Granulomatosis With Polyangiitis (EGPA); Hypereosinophilia Syndrome (HES)
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EGPA/HES Cohort: Benralizumab (Experimental): Participants with greater than or equal to (>=) 35 kg weight will receive benralizumab dose-1 and participants with less than (<) 35 kg weight will receive benralizumab dose-2 as SC injection Q4W during the 52-week treatment period. All participants who complete the 52-week treatment period will be offered the opportunity to continue into an extension period.
  Interventions: Drug: Benralizumab

INTERVENTIONS:
Drug: Benralizumab — Benralizumab will be administered as SC injection on Q4W.
  Other Names: FASENRA

SUMMARY:
The main purpose of study is to assess the safety, tolerability, pharmacokinetics (PK), and efficacy of benralizumab.

DETAILED DESCRIPTION:
This study is open-label, multicentre, basket study to evaluate the safety, PK, pharmacodynamic (PD), efficacy, and immunogenicity of repeat dosing of benralizumab subcutaneous (SC) every 4 weeks (Q4W) in male and female children with rare eosinophilic diseases.

Paediatric participants with eosinophilic granulomatosis with polyangiitis (EGPA) will be enrolled in the first cohort.

Paediatric participants with hypereosinophilic syndrome (HES) will be enrolled in the second cohort. Additional cohorts in other eosinophilic diseases may be added in future protocol amendments.

The study consists of 3 periods:

1. Screening period: 1 to 4 weeks
2. Open-label treatment period: 52 weeks
3. Open-label extension period: at least 52 weeks (plus safety follow-up [SFU] weeks after last investigational product [IP] administration)

All eligible participants will receive benralizumab SC Q4W during the 52-week open-label treatment period.

All participants who complete the 52-week open-label treatment period on IP will be offered the opportunity to continue into an extension period. The extension period is intended to allow each participant at least an additional one year of treatment with benralizumab.

ELIGIBILITY:
Inclusion Criteria:

All Cohorts:

* Male or female participants must be aged 6 to < 18 years of age at the time of signing the assent form and their caregiver signing the informed consent form.
* Body weight greater than (>=) 15 kilograms (kg).

EGPA Cohort:

* Therapy with corticosteroids: The prescribed dose of oral corticosteroids (OCS) (greater than [>] 0.1 milligrams per kilogram per day (mg/kg/day), max dose of 50 milligrams per day (mg/day) must be stable (that is, no adjustment of the dose) for at least 4 weeks prior to baseline (Visit 2).
* Immunosuppressive therapy: If receiving immunosuppressive therapy, the dosage must be stable for at least 4 weeks prior to baseline (Visit 2).

HES Cohort:

* Documented HES diagnosis, defined as history of persistent eosinophilia >1500 cells/µL without secondary cause on 2 examinations ≥1 month apart and evidence of eosinophil-mediated organ involvement.
* Symptomatic active HES, or history of a prior flare, or considered eligible based on disease severity per investigator judgement.
* AEC ≥1000 cells/µL at screening (Visit 1).
* Documented negative testing for Fip1-like 1 gene fused with the platelet-derived growth factor receptor alpha gene (FIP1L1-PDGFR) fusion tyrosine kinase gene translocation.

Exclusion Criteria:

All Cohorts:

* Any current malignancy or history of malignancy.
* History of anaphylaxis to any biologic therapy or vaccine.
* Known, pre-existing, clinically significant endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological, respiratory, or any other system abnormalities.
* Previous receipt of benralizumab in an interventional clinical study.

EGPA Cohort:

* Diagnosed with granulomatosis with polyangiitis (previously known as Wegener'granulomatosis) or microscopic polyangiitis.
* EGPA relapse: any deterioration in EGPA and/or organ-threatening EGPA that per Investigator judgement renders participants unstable in their EGPA within 3 months prior to screening (Visit 1) and through first administration of IP at baseline (Visit 2).
* Life-threatening EGPA: imminently life-threatening EGPA disease within 3 months prior to screening (Visit 1) and through first administration of IP at baseline (Visit 2), as per Investigator judgement.

HES Cohort:

* Life-threatening HES or HES complications, as judged by the investigator.
* Hypereosinophilia of unknown significance (HE-US).
* Diagnosis of systemic mastocytosis.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-10-06 (Estimated); Study Completion 2028-04-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | From screening (Week -4 to -1) until Week 52
  The safety and tolerability of benralizumab will be evaluated.
Serum Concentrations of Benralizumab | Weeks 0, 12, 24, 25, 36, and 52
  The PK of benralizumab will be evaluated.

SECONDARY OUTCOMES:
EGPA Cohort: Percentage of Participants with Remission at Week 24 | At Week 24
  Remission defined as Paediatric Vasculitis Activity Score (PVAS) = 0 and oral corticosteroid (OCS) intake less than or equal to (<=) 0.1 mg/kg/day.
Number of Participants with Positive Antidrug Antibody (ADA) | Weeks 0, 12, 24, 36, 48, and 52
  The immunogenicity of benralizumab will be evaluated.
Change From Baseline in Peripheral Blood Eosinophil Count | From Baseline to Weeks 0, 12, 24, 36, 52
  The PD effect of benralizumab on peripheral blood eosinophil count will be evaluated.
EGPA Cohort: Time to First EGPA Relapse | Up to 52 weeks
  The efficacy of benralizumab on time to first relapse will be assessed. EGPA relapse will be defined as worsening or persistence of active disease since the last visit characterized by: a) Active vasculitis (PVAS > 0); OR b) Worsening of asthma symptoms (based on Asthma Control Questionnaire - Interviewer Administered [ACQ-IA]); OR c) Active nasal and/or sinus disease with worsening in at least one sino-nasal symptom question warranting any of the following: 1) Increase OCS; OR 2) Increase/addition of immunosuppressive medication; OR 3) Hospitalisation related to EGPA worsening.
HES Cohort: Time to first HES worsening/flare | Up to 52 weeks
  The effect of benralizumab on HES worsening/flares will be evaluated.
HES Cohort: Percentage of participants who experience a HES worsening/flare | Up to 52 weeks
  The effect of benralizumab on HES worsening/flares will be evaluated.
HES Cohort: Number of HES worsening/flares (annualised rate/year) | Up to 52 weeks
  The effect of benralizumab on HES worsening/flares will be evaluated. The annualised HES worsening/flare rate will be calculated as follows:
  The total number of flares *365.25 / total duration of follow-up in the treatment period (days).
HES Cohort: Percentage of Participants requiring an increase in corticosteroid dose | Up to 52 weeks
  The effect of benralizumab on corticosteroid use will be evaluated.
HES Cohort: Time to first haematologic relapse | Up to 52 weeks
  The time to first haematologic relapse will be defined as the time from first dose of IP to the first post baseline visit with Absolute eosinophil count [AEC] ≥ 1000 cells/uL.
HES Cohort: Percentage of Participants with haematologic relapse | Up to 52 weeks
  The effect of benralizumab on haematologic measures of disease activity will be evaluated.
HES Cohort: Percentage of Participants who have AEC < 500 cells/μL for 24 weeks | Up to 52 weeks
  The effect of benralizumab on haematologic measures of disease activity will be evaluated.
HES Cohort: Patient Global Impression of Change (PGI-C) Score | Weeks 12, 24, 36 and 48
  The effect of benralizumab on participant/caregiver reported measures of disease severity and health status will be assessed. The PGI-C instrument captures the participant's overall evaluation of response to treatment, and rated on a 7-point PGI-C scale ranging from 1 ('much better') to 7 ('much worse').

CONTACTS AND LOCATIONS:
Locations (6):
- Research Site, Aurora, Colorado, United States
- Research Site, São Paulo, Brazil
- Research Site, Toronto, Ontario, Canada
- Research Site, Guadalajara, Mexico
- Turkey (Türkiye) (2):
  - Research Site, Altındağ
  - Research Site, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via there quest portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment athttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/